CLINICAL TRIAL: NCT00830778
Title: Reduced Postoperative Pancreatic Fistula Rate Following Pancreaticoduodenectomy; Multicentric Randomized Controlled Trial on Pancreaticogastrostomy vs. Pancreaticojejunostomy
Brief Title: Reduced Pancreatic Fistula Rate Following Pancreaticoduodenectomy: Trial on Pancreaticogastrostomy Versus Pancreaticojejunostomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baki Topal (Other)
Collaborators: Erasme ULB, Brussels (Unknown); Jolimont, Brussels (Unknown); St.Lucas, Brugge (Unknown); General Hospital Groeninge (Other); Université Catholique de Louvain (Other); Clinique Saint Joseph, Liège (Other); University Hospital, Antwerp (Other); Jan Palfijn, Antwerp (Unknown); AZ Sint-Lucas Brugge (Other); Monica, Deurne (Unknown)
Responsible Party: Sponsor-Investigator, Baki Topal, MD, PhD, University Hospital, Gasthuisberg
Organization: University Hospital, Gasthuisberg (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: S51480
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Tumors
Keywords: pancreas; surgery; cancer; pancreaticoduodenectomy (PD); peri-ampullary tumours (ampulla, duodenum, distal bile duct, and miscellaneous tumours); pancreatic tumors; peri-ampullary tumors
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms | interventions — Pancreaticojejunostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PG anastomosis (Experimental): Pancreaticogastrostomy (PG) reconstruction/anastomosis after pancreaticoduodenectomy (PD)
  Interventions: Procedure: Pancreaticogastrostomy
- PJ anastomosis (Active Comparator): Pancreaticojejunostomy (PJ) reconstruction/anastomosis after pancreaticoduodenectomy (PD)
  Interventions: Procedure: Pancreaticojejunostomy

INTERVENTIONS:
Procedure: Pancreaticojejunostomy — Pancreaticojejunostomy (PJ) reconstruction/anastomosis
  Arms: PJ anastomosis
Procedure: Pancreaticogastrostomy — Pancreaticogastrostomy (PG) reconstruction/anastomosis
  Arms: PG anastomosis

SUMMARY:
The incidence of complications after pancreaticoduodenectomy (PD) is around 50 %. The postoperative course after PD is strongly dependent of the occurrence of pancreatic fistula (POPF), which determines postoperative mortality, length of hospital stay and costs. The incidence of POPF after PD is dependent of its definition, and is reported in up to 20% of patients.

There is disagreement on whether to perform a pancreaticojejunostomy (PJ) or a pancreaticogastrostomy (PG) after PD. The aim of the current randomized controlled trial is to study whether PG significantly reduces the rate of POPF following PD for pancreatic or peri-ampullary tumours. Secondary endpoints are the reduction of overall postoperative complication rate and their severity.

DETAILED DESCRIPTION:
Therapeutic intervention

* Surgeons who have performed a minimum of five (5) PG and PJ procedures can include patients in this randomized trial.
* Any dissection device or technique is allowed.
* Pancreatic anastomosis (PG or PJ)

  * 1-layer or 2-layer anastomosis is allowed but has to be registered
  * mono-filament and/or poly-filament suture material is allowed but has to be registered
  * no pancreatic stent will be placed
* Drainage: one (1) or more closed drain(s) with or without suction is allowed in the vicinity of the pancreatic anastomosis
* Enteral tube feeding (tube positioned in the jejunum at the time of surgery, and distal to the pancreatic anastomosis) as well as total parenteral nutrition (TPN) is allowed
* Gastrostomy tube (percutaneous) is allowed
* Somatostatin: start intra-operatively and administered for seven (7) days after surgery at a dose of 6 mg/d
* Prophylactic use of antibiotics during 24h post-operatively
* Prophylactic use of Ranitidine as well as any PPI (proton pump inhibitor) is allowed to prevent peptic ulcer

Clinical evaluation and assessment criteria

* The number and type of POPF will be recorded according to the ISGPF guidelines and based on findings on day 3 (three) after surgery
* The number and type of postoperative complications will be recorded. The therapy-oriented severity grading system (TOSGS) of complications will be used and complications will be allocated to surgical (SSC) and non-surgical site (NSSC) complications
* The adequacy of the surgical resection margins (pR0) and the magnitude of the tumour-free resection margin (millimetres) will be monitored
* Postoperative length of hospital stay (LOS) will be registered

Patient randomization and registration procedure (randomization lists attached)

* This is a multicentric randomized controlled trial.
* Patient randomization will be done intra-operatively since a substantial number of patients could be dropped out intra-operatively because of the presence of unexpected intra-abdominal metastases at the time of surgery.
* Patient stratification will be performed for each centre and will be based on the diameter of the pancreatic duct. A pancreatic duct at the level of the surgical transsection margin measuring 3 millimetres or less in diameter is defined as being a "soft pancreas". A pancreatic duct measuring more than 3 millimetres is defined as a "hard pancreas".
* A prospective registration of following parameters will be performed: intra-operative diameter of the pancreatic duct at the surgical transection margin, diameter of the pancreas at the surgical transection margin, pancreatic tissue consistency assessed by the surgeon: soft vs. hard, post-operative pathology parameters.

Statistical analysis and sample size calculation based on a stratified design

* 40% of patients are expected to have a hard pancreas and 60% a soft pancreas.
* It is assumed that the magnitude of the effect of the intervention (PJ vs. PG) on the POPF rate, expressed as an odds ratio (OR), is similar in both strata.
* The needed sample size is calculated to have 80% power to detect a common odds ratio of 2.7. POPF rates of 12% and 20% are assumed after PJ within the hard and soft pancreas stratum respectively (yielding 4.8% and 8.4% after PG). Note that, given the unequal size strata, this leads to an expected POPF rate of 16.8% after PJ and 7% after PG (≈12% POPF overall).
* A 2-sided (with alpha=5%) Mantel-Haenszel test of OR=1 for stratified 2x2 tables is planned
* 168 patients are required per group (total patient population 336)
* Expected duration of recruitment: 3-4 years
* An interim analysis will be performed annually (i.e. after inclusion of 1/3 and 2/3 of the patients) to to allow early stop of the study (or accrual of patients in a specific treatment group) due to rejection of the null hypothesis. Using the O'Brien-Fleming method (O'Brien and Fleming 1979) results in respectively |3.471|, |2.454| and |2.004| as critical values for the Z-statistic at the three analysis moments. Otherwise stated, p-values are declared significant if <.00052, <0.0141 and <0.0451 at respectively the first interim analysis, the second interim analysis and at the final analysis.
* Exact 95% confidence intervals will be calculated for the POPF and post-operative complication rates within each stratum. A stratified Mann-Whitney U test will be used for the TOSGS grading.

Translational research: optional Prognostic relevance of gene expression profiling in pancreatic cancer: analyses will be performed at UZ.Leuven/KU.Leuven (project coordinator B.Topal)

* Fresh tissue samples from pancreatic cancer and from non-tumoral pancreatic tissue will be stored in RNA-later (samples in 2 separate tubes; 5-10 volumes of RNA-later)
* Sample tubes will be transported (or picked up by the coördinator's research team), within 3 days from sampling, to be stored in -80°C for further analyses

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, who undergo PD for a pancreatic or peri-ampullary tumor
* Age between 18 to 85 years
* Patients with and without pre-operative biliary drainage (for obstructive jaundice)
* Concomitant surgical procedures such as simultaneous colonic resection etc.
* Reconstruction of the portal vein or superior mesenteric vein

Exclusion Criteria:

* Age < 18years
* Pregnancy
* Pre-operative radiotherapy
* PD for IPMT
* PD for chronic pancreatitis
* PD for pancreatic trauma
* PD for post-ERCP complications
* Any arterial reconstruction at the time of surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Reduction of clinical postoperative pancreatic fistula (POPF) rate | 3 years

SECONDARY OUTCOMES:
Reduction of overall postoperative pancreatic fistula rate | 3 years
Reduction of the severity of postoperative complications | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Baki Topal, MD, PhD, Study Director — Universitaire Ziekenhuizen KU Leuven; Claude Bertrand, MD, Principal Investigator — Hospital Jolimont, Brussels; Jean Closset, MD, PhD, Principal Investigator — Hospital Erasme (ULB), Brussels; Henk Thieren, MD, Principal Investigator — AZ. St.Lucas, Brugge; Franky Vansteenkiste, MD, Principal Investigator — General Hospital Groeninge; Jean-Francois Gigot, MD, PhD, Principal Investigator — Université Catholique de Louvain; Joseph Weerts, MD, Principal Investigator — St.Joseph Hospital, Liège; Geert Roeyen, MD, Principal Investigator — University Hospital Antwerp, Antwerp; Marc Janssens, MD, Principal Investigator — J.Palfijn Hospital, Antwerp; Tom Feryn, MD, Principal Investigator — St.Jan Hospital, Brugge; Steven Pauli, MD, Principal Investigator — Monica Hospital, Deurne
Locations (1):
- University Hospital Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Derived] Topal B, Fieuws S, Aerts R, Weerts J, Feryn T, Roeyen G, Bertrand C, Hubert C, Janssens M, Closset J; Belgian Section of Hepatobiliary and Pancreatic Surgery. Pancreaticojejunostomy versus pancreaticogastrostomy reconstruction after pancreaticoduodenectomy for pancreatic or periampullary tumours: a multicentre randomised trial. Lancet Oncol. 2013 Jun;14(7):655-62. doi: 10.1016/S1470-2045(13)70126-8. Epub 2013 May 2. PMID 23643139
- [Derived] Bertrand C, Squifflet JP, Gys T, Berrevoet F, Jehaes C, Lerut T, Malaise J, Topal B. The Society for Internet-based Scientific Studies: a new platform to promote multicentric studies in the Royal Belgian Society for Surgery. Acta Chir Belg. 2010 Jan-Feb;110(1):3-5. doi: 10.1080/00015458.2010.11680554. No abstract available. PMID 20306901